CLINICAL TRIAL: NCT00799968
Title: Efficacy and Safety Evaluation of 12-h and 2-h Urokinase Regimes in the Treatment of Pulmonary Thromboembolism: A Multi-Center, Randomized Controlled Trial in China
Brief Title: 12-h and 2-h Urokinase Regimes of Pulmonary Thromboembolism in China
Acronym: UKPTEC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Beijing Chao Yang Hospital, Chen WANG,Beijing Institute of Respiratory Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004BA703B07-UK
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Pulmonary Embolism; Thromboembolism
Keywords: Thrombolytic therapy; Urokinase; Efficacy; Safety
MeSH Terms: conditions — Pulmonary Embolism; Thromboembolism | interventions — Urokinase-Type Plasminogen Activator; Fibrinolytic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): UK-12h group
  Interventions: Drug: Urokinase
- Group 2 (Experimental): UK-2h group
  Interventions: Drug: Urokinase

INTERVENTIONS:
Drug: Urokinase — UK,bolus 4 400 U/kg followed by intravenous 2 200 U/kg•h for 12 hours
  Other Names: Urokinase,thrombolytic agent
  Arms: Group 1
Drug: Urokinase — UK,20 000U/kg continuously intravenous infusion for 2 hours
  Other Names: Urokinase,thrombolytic agent
  Arms: Group 2

SUMMARY:
Comparative trials of urokinase (UK) for 12 hours（UK-12h）or 24 hours (UK-24h) have produced similar results in acute pulmonary thromboembolism (PTE) thrombolysis. It is unclear whether the infusion time can be reduced further. The aim of this study was to investigate the efficacy and safety of weight adjusted dosage of UK-2h (20 000 IU/Kg) regime with the Uk-12h regime in selected patients with PTE in Chinese population.

DETAILED DESCRIPTION:
Pulmonary thromboembolism (PTE), a frequent life-threatening complication of deep vein thrombosis (DVT), is often underestimated and under diagnosed . Effective early treatment will decrease the mortality, reverse right heart dysfunction and reduce risk of chronic thromboembolic pulmonary hypertension (CTEPH) or post-thrombotic syndrome (PTS). Thrombolysis has proved to be the most rapid and effective therapy to reduce the obstruction of pulmonary circulation and normalize hemodynamic parameters. The ultimate goals of thombolytic therapy for this disease are to minimize early morbidity and mortality and to prevent recurrence without provoking excessive bleeding.

Currently, the choice of thrombolytic agents and regimens (either UK or rt-PA) is mostly based on personal or regional preferences. A loading dose of UK 4400 IU/kg followed by 2200 IU/kg/hour for 12 hours (UK-12h), or rt-PA 100 mg infusion over 2 hours are recommended for acute PTE treatment. However, increasing evidence suggest that UK infusion can be more concentrated and time can be further reduced. 100 mg/2 h of rt-PA and a novel dosing regimen of UK(3 million U/2 h) had been compared. The results indicated that a 2-h regimen of rt-PA and 2h UK exhibited similar efficacy and safety for treatment of acute PTE. UK-2h(20 000U/Kg) regimen combined with low molecular weight heparin (LMWH) had been used in Chinese population.No severe bleeding and allergic reaction occurred in the thrombolytic group. This dosage is much lower than that used by Goldhaber et al, but the efficacy was prominent. Until now,no study have been reported to compared UK-2h(20 000U/Kg) regimen with other UK regimens(such as UK-12h).

A relative lower dosage of UK 2-h regimen with body weight adjusted may be an alternative choice for treating PTE patients in Chinese population.Considering lower cost and convenience of this regimen, the efficacy and safety between UK-2h regimen(20 000U/Kg) and ACCP-approved UK-12h regimen for treating acute PTE will be compared.The study is conducted on patients with massive PTE with shock or hypotension and/or if without shock or hypotension but with right ventricular dysfunction. The clinical efficacy, emboli dissolving efficacy and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* PTE confirmed either by a high probability ventilation-perfusion lung scanning (V/Q scan) or by CTPA.
* massive PTE patients with haemodynamic instability and/or cardiogenic shock
* Anatomic obstruction more than 2 lobes on CTPA and/or defect more than 7 segments on V/Q scan with evidence of right ventricular dysfunction (RVD) and pulmonary hypertension on echocardiography
* Symptoms within 15 days
* Written informed consent was obtained from all the patients before randomization

Exclusion Criteria:

* Received parenteral heparin for more than 72 hours
* Known allergic to urokinase
* Thrombolytic contraindications such as:

  1. active bleeding or spontaneous intracranial hemorrhage;
  2. major surgery, organ biopsy or recent puncture of a non-compressible vessel less than 10 days;
  3. cerebral arterial thrombosis within 2 months;
  4. gastro-intestinal bleeding within 10 days;
  5. major trauma within the past 15 days;
  6. neurosurgery or ophthalmologic operation with 30 days;
  7. uncontrolled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg);
  8. recent external cardiac resuscitation manoeuvres;
  9. platelet count < 100 000/mm3 at admission;
  10. pregnancy, puerperium or lactation with 2 weeks;
  11. infectious pericarditis or endocarditis;
  12. severe hepatic and kidney dysfunction;
  13. hemorrhagic retinopathy due to diabetes;
  14. a known bleeding disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2002-06; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The improvement of the right ventricular function , perfusion defect score on lung V/Q scans or quantitative computed tomographic pulmonary angiography (CTPA) score. | 14d

SECONDARY OUTCOMES:
The incidence of major or minor bleeding, death rate, and PTE recurrence at 14d after treatment. | 14d

CONTACTS AND LOCATIONS:
Overall Officials: Chen WANG, Prof, Principal Investigator — Beijing Institute of Respiratory Medicine,Beijing Chao Yang Hospital
Locations (31):
- China (31):
  - Beijing Chaoyang Hospital, Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Beijing General Hospital of the Air-force PLA, Beijing, Beijing Municipality
  - Beijing Fu Xing Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Naval General Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital Sun Yat-Sen University, Guangzhou, Guandong
  - Guangzhou Institute of Respiratory Disease，Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan Worker's Hospital, Hebei Medical University, Tangshan, Hebei
  - The Affiliated Hospital of Hubei Coal University, Tangshan, Hebei
  - Wuhan Union Hospital, Wuhan, Hubei
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The General Hospital of Shenyang Military Command, Shenyang, Liaoning
  - Qilu Hospital Affiliated to Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Medical College Qingdao, Qingdao, Shandong
  - Shangdong Yantaishan Hospital, Yantai, Shandong
  - The First Affiliated Hospital of Jining Medical College, Jinan, Shangdong
  - The First Affiliated Hospital of Qingdao University CHENG Zhao-zhong, Qingdao, Shangdong
  - The Fifth People's Hospital of Datong in ShanxiWANG;, Datong, Shanxi
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin Thoracic Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Xinjiang People's Hospital, Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital, Affiliated with Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang

REFERENCES:
- [Background] Pang BS, Wang C, Lu Y, Yang YH, Xing GH, Mao YL, Huang XX, Zhai ZG. [Changes of blood coagulative and fibrinolytic system and function of pulmonary vascular endothelium after therapy in patients with acute pulmonary thromboembolism]. Zhonghua Yi Xue Za Zhi. 2007 Nov 20;87(43):3074-8. Chinese. PMID 18261355
- [Background] Zhu L, Yang Y, Wu Y, Zhai Z, Wang C. Value of right ventricular dysfunction for prognosis in pulmonary embolism. Int J Cardiol. 2008 Jun 23;127(1):40-5. doi: 10.1016/j.ijcard.2007.06.093. Epub 2007 Aug 22. PMID 17716753
- [Background] Liu Y, Wang C, Yang Y, Hou X, Wang J. Pro-urokinase up-regulates the expression of urokinase-type plasminogen activator (u-PA) in human pulmonary arterial endothelial cells. Thromb Res. 2008;121(4):485-91. doi: 10.1016/j.thromres.2007.05.021. Epub 2007 Jul 20. PMID 17640719
- [Background] Zhu L, Wang C, Yang Y, Wu Y, Zhai Z, Dai H, Pang B, Tong Z. Value of transthoracic echocardiography in therapy regimens evaluation in pulmonary embolism. J Thromb Thrombolysis. 2008 Dec;26(3):251-6. doi: 10.1007/s11239-007-0087-8. Epub 2007 Aug 21. PMID 17705052
- [Background] Zhu L, Yang YH, Wu YF, Zhai ZG, Wang C; National Project of the Diagnosis and Treatment Strategies for Pulmonary Thromboembolism investigators. Value of transthoracic echocardiography combined with cardiac troponin I in risk stratification in acute pulmonary thromboembolism. Chin Med J (Engl). 2007 Jan 5;120(1):17-21. PMID 17254482
- [Background] Zhai ZG, Wang C, Yang YH, Pang BS, Xiao B, Liu YM, Mao YL, Weng XZ. [Relationship between polymorphisms of plasminogen activator inhibitor-1 promoter gene and pulmonary thromboembolism in Chinese Han population]. Zhonghua Yi Xue Za Zhi. 2006 May 23;86(19):1313-7. Chinese. PMID 16796899
- [Background] Liu CP, Zhang YJ, Lu WX, Ji YQ, Zhang WH, Wang C. [The change of pulmonary surfactant associated protein A in acute pulmonary embolism]. Zhonghua Jie He He Hu Xi Za Zhi. 2005 Sep;28(9):600-3. Chinese. PMID 16207426
- [Background] Ren H, Su PX, Zhang CJ, Gu S, Ma GT, Zhang H, Wang C. [Surgical treatment of chronic pulmonary thromboembolism]. Zhonghua Wai Ke Za Zhi. 2005 Mar 15;43(6):345-7. Chinese. PMID 15854334
- [Background] Wang C, Cheng XS, Zhong NS. [Promoting the clinical and research work on pulmonary thromboembolism in China]. Zhonghua Jie He He Hu Xi Za Zhi. 2004 Nov;27(11):721-2. No abstract available. Chinese. PMID 15634378
- [Background] Pang BS, Wang C, Luo Q, Zhang LM, Zhu M, Mao YL, Huang XX, Guo WJ. [Study of the function of coagulation, fibrinolysis and pulmonary vascular endothelium before and after experimental pulmonary thromboembolism in rabbits]. Zhonghua Jie He He Hu Xi Za Zhi. 2004 Jun;27(6):381-4. Chinese. PMID 15256085
- [Background] Wang F, Wang C, Wang T, Pang BS, Wu YB, Yang YH, Li C, Zhang HY, Weng XZ. [Experimental study of the thrombolytic effects in a canine model of pulmonary thromboembolism induced by autologous radioactive blood clots]. Zhonghua Jie He He Hu Xi Za Zhi. 2004 Feb;27(2):93-6. Chinese. PMID 14990182
- [Background] Zai ZG, Wang C. [Advances in the study of pulmonary thromboembolism]. Zhonghua Jie He He Hu Xi Za Zhi. 2004 Jan;27(1):14-8. No abstract available. Chinese. PMID 14989818
- [Background] Qin ZQ, Wang C. [Comparison of thrombolysis and anticoagulation in pulmonary thromboembolism: a meta-analysis]. Zhonghua Jie He He Hu Xi Za Zhi. 2003 Dec;26(12):772-5. Chinese. PMID 14720434
- [Background] Wang F, Wang C, Wang T, Pang BS, Wu YB, Yang YH, Li C, Zhang HY, Weng XZ. [A canine model of acute pulmonary thromboembolism induced by autologous radioactive blood clots]. Zhonghua Jie He He Hu Xi Za Zhi. 2003 Aug;26(8):470-3. Chinese. PMID 14505523
- [Derived] Wang C, Zhai Z, Yang Y, Yuan Y, Cheng Z, Liang L, Dai H, Huang K, Lu W, Zhang Z, Cheng X, Shen YH; China Venous Thromboembolism Study Group. Efficacy and safety of 2-hour urokinase regime in acute pulmonary embolism: a randomized controlled trial. Respir Res. 2009 Dec 29;10(1):128. doi: 10.1186/1465-9921-10-128. PMID 20040086